CLINICAL TRIAL: NCT05446779
Title: Postmortem Evaluation of Adrenal and Other Endocrine Tumors in Patients With Sudden Death Without Definitive Causative Diagnosis (PEA-SuddenDeath)
Brief Title: Postmortem Evaluation of Adrenal and Other Endocrine Tumors in Patients With Sudden Death
Acronym: SuddenDeath
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); University of Helsinki (Other); Tampere University Hospital (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Niina Matikainen, M.D., Ph.D, , Assoc. Prof., Helsinki University Central Hospital
Other Study IDs: THL/5008/5.05.00/2021
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Primary Aldosteronism; Adrenal Cushing Syndrome; Pheochromocytoma; Endocrine Neoplasia
MeSH Terms: conditions — Hyperaldosteronism; ACTH Syndrome, Ectopic; Pheochromocytoma; Endocrine Gland Neoplasms | interventions — Staining and Labeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sudden death: Unexpected witnessed death occurring within an hour of the onset of symptoms in a person with or without previously known cardiac disease without an extra-cardiac cause, or unexpected unwitnessed death without extra-cardiac cause occurring in the previous 24 hours
  Interventions: Diagnostic Test: Adrenal aldosterone synthase (CYP11B2) staining; Diagnostic Test: Adrenal cortisol synthase (CYP11B1) staining; Diagnostic Test: Histopathological analysis
- Control: Death because of an exogenic reason for sudden death such as trauma or suicide as a control group i.e. non-disease-induced sudden death
  Interventions: Diagnostic Test: Adrenal aldosterone synthase (CYP11B2) staining; Diagnostic Test: Adrenal cortisol synthase (CYP11B1) staining; Diagnostic Test: Histopathological analysis

INTERVENTIONS:
Diagnostic Test: Adrenal aldosterone synthase (CYP11B2) staining — Immunoshistochemical diagnosis of primary aldosteronism
Diagnostic Test: Adrenal cortisol synthase (CYP11B1) staining — Immunoshistochemical diagnosis of adrenal hypercortisolism
Diagnostic Test: Histopathological analysis — Diagnosis of any endocrine neoplasia other than primary aldosteronism or adrenal hypercortisolism

SUMMARY:
Sudden Cardiac Death is a leading cause of mortality and remains a major public health burden worldwide. Cardiac arrest due to coronary heart disease explains a large proportion of the cases, but if autopsy is not performed the exact underlying cause remains obscure in many adults who face sudden death outside heath care organizations. The investigators aim to find proof that primary aldosteronism is a risk factor for sudden death and to characterize the prevalence of adrenal pathology in sudden death of undetermined cause in a case-control study. In addition, the study aims to characterize the prevalence of other adrenal pathology i.e. silent adenomas, cortisol-producing adenomas and pheochromocytomas in sudden death. The investigators also seek evidence that other endocrine hormone overproduction-causing diseases are more prevalent in persons with sudden death compared with those experiencing traumatic or suicidal death sudden death.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients with out-of-hospital, sudden death

Exclusion Criteria:

1. Estimated time from death to refrigerator more than 24-48 hours and in the refrigerator time more than 7 days (susceptibility to excessive tissue breakdown)
2. Terminal disease
3. Institutionalized patients

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enroll aproximately 200 consecutive patients with out-of-hospital, sudden death to both groups.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CYP11B2 staining in adrenal glands | Through study completion, an average of 2 years
  Histopathological diagnosis of the autopsy
CYP11B1 staining in adrenal glands | Through study completion, an average of 2 years
  Histopathological diagnosis of the autopsy

SECONDARY OUTCOMES:
CYP11B2 staining in adrenal glands | Through study completion, an average of 2 years
  Histopathological diagnosis of the autopsy
Pheochromocytoma or paraganglioma | Through study completion, an average of 2 years
  Histopathological diagnosis of the autopsy
Neuroendocrine tumor | Through study completion, an average of 2 years
  Histopathological diagnosis of the autopsy

CONTACTS AND LOCATIONS:
Overall Officials: Niina Matikainen, MD, PhD, Assoc Prof, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Endocrinology, Helsinki University Hospital and University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ylanen A, Isojarvi J, Virtanen A, Leijon H, Vesterinen T, Aro AL, Huhtala H, Kokko E, Porsti I, Viukari M, Nevalainen PI, Matikainen N. Adrenal aldosterone synthase (CYP11B2) histopathology and its association with disease-induced sudden death: a cross-sectional study. Lancet Reg Health Eur. 2025 Feb 6;51:101226. doi: 10.1016/j.lanepe.2025.101226. eCollection 2025 Apr. PMID 39995489